CLINICAL TRIAL: NCT04761575
Title: Validation and Reproducibility Study of the eNutri Online Food Frequency Questionnaire for UK Adults Aged 65 Years and Older
Brief Title: Validation of the eNutri Food Frequency Questionnaire for Adults Aged 65 y and Older
Acronym: eNutriFFQ65+
Status: Completed | Type: Observational
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Julie Lovegrove, Director of the Hugh Sinclair Unit of Human Nutrition, University of Reading
Other Study IDs: 20/40
Record Dates: First submitted 2021-02-12; First posted 2021-02-21 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Diet Habit
Keywords: Food frequency questionnaire; Nutrition; Dietary intake
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Dried blood spots will be collected from participants but will not be used to extract DNA. The dried blood spots will be used to validate the FFQ against selected biomarkers such as markers of health (e.g. cholesterol) and markers of nutrient intake (e.g. carotenoids).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FFQ validation: All participants to complete all aspects of the study.
  Interventions: Other: Validation of the FFQ65+ via eNutri app

INTERVENTIONS:
Other: Validation of the FFQ65+ via eNutri app — All participants will provide two eNutri FFQ datasets within a 14-day interval along with three 24-hour dietary recalls and dried blood spot samples.

SUMMARY:
The aim is to determine whether the eNutri web application can effectively estimate the dietary intake of a UK older population. The eNutri FFQ65+ study will validate the eNutri online food frequency questionnaire (FFQ) using 100 adults aged 65+ years. The FFQ will be validated against an online 24-hour dietary recall system (Intake24) and its reproducibility will be evaluated by the completion of two FFQs within a 14-day interval. In addition, all participants will also be asked to provide dried blood spot (DBS) samples which will be analysed for key biomarkers of nutritional intake and health. Biomarker results will be compared to FFQ results to further validate the eNutri FFQ.

DETAILED DESCRIPTION:
The primary objective of this study is to validate the eNutri FFQ65+ that assesses dietary intake for the previous 4 weeks against a widely-used, validated computer based 24-hour dietary recall system (Intake24), which is the dietary assessment tool currently used by the UK's National Diet and Nutrition Survey Rolling Programme. The second objective, the reproducibility of the FFQ 65+ dietary data, will also be tested by asking participants to complete the eNutri FFQ on two separate occasions with a 14-day interval between both. In addition, after completing the first FFQ, DBS will be collected from all participants to further validate the FFQ results against selected biomarkers, for example markers of nutrient intake, such as carotenoids, and markers of health, such as cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 years or over
* Live in the UK
* Able to spend approximately 30 minutes using a screen on a device
* Do not have a diagnosis of dementia or another condition affecting memory
* Do not have a food allergy or food intolerance (self- or medically diagnosed)
* Are not following a weight loss diet
* Generally eat on 2 or more occasions everyday

Exclusion Criteria:

* Follow a specialised or restricted diet (not including vegan and vegetarian diets)
* Have a medical condition or take medications that do not allow an individual to eat a stable diet on a day-to-day basis (e.g. severe gastrointestinal condition)
* Anticipate changes to their diet within the next three weeks (e.g. surgery, holiday, receiving nutritional advice from a professional)
* Have participated in another nutrition study that included a specific dietary regime in the last 4 weeks or are currently participating

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Adults aged 65 and over who live in the UK
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
eNutri dietary intake | Baseline
  eNutri FFQ1 dietary data

SECONDARY OUTCOMES:
eNutri dietary intake | Day 14
  eNutri FFQ2 dietary data

OTHER OUTCOMES:
24-hour dietary recall intake | Baseline
  Self-reported 24-hour dietary intake using Intake24 on three randomly allocated days within 14 days
Dried blood spot biomarkers | Baseline
  Dried blood spots analysed for selected biomarkers such as markers of health (e.g. cholesterol) and dietary intake (e.g. carotenoids).
Height | Baseline
  Self-reported measurement of height
Weight | Baseline
  Self-reported measurement of weight
Weight | Day 14
  Self-reported measurement of weight

CONTACTS AND LOCATIONS:
Overall Officials: Julie Lovegrove, Professor, Principal Investigator — Hugh Sinclair Unit of Human Nutrition, University of Reading
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The researchers are part of the FNS-Cloud Consortium. Anonymised FFQ, 24h recall and DBS data will be on shared on FNS-Cloud (in development; https://www.fns-cloud.eu/) at the end of the project.
Time Frame: Data available at the end of the project.
Access Criteria: Will depend on FNS-Cloud access criteria (https://www.fns-cloud.eu/) - to be decided by the consortium.